CLINICAL TRIAL: NCT06266780
Title: Impact Evaluation of a Targeted mHealth Intervention to Improve Uptake of Postpartum Contraception in Kenya
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacaranda Health (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Jhpiego (Other); IPSOS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: P1473-2023
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Family Planning
Keywords: Maternal Health; Postpartum Health; Contraception; Family Planning; Birth Spacing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Group receiving enhanced package of postpartum family planning support
  Interventions: Behavioral: PROMPTS Enhanced Family Planning Counselling
- Control Group (No Intervention): Group receiving basic postpartum family planning information

INTERVENTIONS:
Behavioral: PROMPTS Enhanced Family Planning Counselling — Based on a targeted human-centered-design process with pregnant and early postpartum mothers, the intervention consists of informative messages, counselling and reminders regarding postpartum family planning and birth spacing, leveraging an existing mobile health platform (PROMPTS) for intervention delivery and Jacaranda's established partnership with the Kenyan Ministry of Health, county health offices and public maternity hospitals method options. The intervention includes several features: activation of family planning discussions between pregnant and postpartum women and their health care providers, information provision, method selection support to help women choose their preferred method, and reminders to follow-up. The key feature is to help women make an informed plan about family planning in the prenatal or early postpartum period and follow through with this plan.
  Arms: Intervention Group

SUMMARY:
The goal of this study is to explore approaches to improve postpartum contraceptive counseling, information, and uptake through a collaboration between the Harvard Chan School, Rutgers School of Public Health, Jacaranda Health, Jhpiego, and IPSOS, leveraging an existing mobile health platform for intervention delivery and Jacaranda's established partnership with the Kenyan Ministry of Health, county health offices and public maternity hospitals.

Jacaranda's PROMPTS mHealth platform has reached over two million pregnant women and new mothers, providing them with needed, tailored information about prenatal and postpartum health along with access to a mobile helpdesk to triage users' questions. Using a targeted human-centered-design process with early postpartum mothers, we developed targeted messaging around family planning and contraceptive method options, with the goal of integrating this new content into Jacaranda's PROMPTS platform. We will conduct a randomized controlled trial with pregnant women engaged with the PROMPTS platform to determine the impact of the intervention package on information and utilization of postpartum contraception. If proven effective, the results of this intervention will be integrated into Jacaranda's PROMPTS system at full scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 and over,
* Pregnant at 7-8 months gestation,
* Consented to be enrolled in the PROMPTS text-messaging platform and who have provided informed consent to be part of this research study
* Have access to a mobile phone

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4190 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of postpartum family planning at 3 months | 3 months
  The outcome is a binary variable, set to 1 if a participant reports using any modern family planning method (including Lactational Amenorrhea Method (LAM)) at the time of the survey. The modern methods considered will include sterilization (both male and female), implants, Intrauterine Device (IUD), injectables, oral contraceptives (pill), condoms (both male and female), diaphragm, foam/jelly, and LAM.
Use of postpartum family planning at 6 months | 6.5 months
  The outcome is a binary variable, assigned a value of 1 if a participant reports using any modern family planning method, excluding LAM, at the time of the survey. The modern methods considered include sterilization (both male and female), implant, IUD, injectables, oral contraceptives (pill), condoms (both male and female), diaphragm, foam, and jelly.

SECONDARY OUTCOMES:
Knowledge of return to fertility | 3 months postpartum
  The outcome is a binary variable, set to 1 if a participant is aware of the possibility of becoming pregnant after giving birth, even if she has not yet seen her period
Knowledge of safe birth spacing | 3 months postpartum
  The outcome is a binary variable, set to 1 if a participant is aware of the minimum recommended delay between the delivery of a baby and the start of the next pregnancy (two years) to promote the health of both the mother and the child.
Knowledge of lactational amenorrhea (LAM) method | 3 months postpartum
  This outcome is an index assessing knowledge of LAM as a method to avoid or delay pregnancy and consists of three items. The first item is a binary indicator, set to 1 if a participant has any familiarity with LAM. The second item is a binary variable, set to 1 if the participant, among those familiar with LAM, knows the recommended duration of LAM use post-delivery (up to 6 months after delivery). The third item is a binary variable, set to 1 if the participant, again among those familiar with LAM, is aware of the other two factors that can reduce the effectiveness of LAM (return of menstruation and the introduction of liquids/foods to the baby). Participants who are not familiar with LAM will automatically receive a score of 0 for the second and third items.
Intention to continue family planning method | 3 and 6.5 months postpartum
  The outcome is a binary variable, assigned a value of 1 if a participant reports an intention to continue using the same family planning method that they were using at the time of the survey.
Intended duration of continued family planning method use | 3 and 6.5 months postpartum
  Among participants who reported an intention to continue with their current family planning method, this outcome quantifies the number of months they plan to maintain its use, as indicated during the survey.
Desired pregnancy spacing of two years or more | 3 months postpartum
  This outcome assesses participants' intentions regarding birth spacing following their recent pregnancy. The primary focus is to determine the proportion of participants planning a gap of at least two years before the onset of their next pregnancy. Participants' intentions are categorized into:
  * Less than 6 months
  * 6 months to less than 12 months
  * 1 year to less than 2 years
  * 2 years or more (main outcome of interest).
Short interpregnancy interval | 3 and 6.5 months postpartum
  The outcome is a binary variable, assigned a value of 1 if a participant reports being pregnant at either of the two follow-up surveys conducted at 3 months or 6.5 months.
Method satisfaction | 3 and 6.5 months postpartum
  This outcome is a discrete variable with values ranging from 1 (very unsatisfied) to 5 (very satisfied), assessing overall satisfaction with the current family planning method. It is evaluated only among participants who reported using a family planning method at the time of the survey.
Uptake of most effective family planning methods | 3 and 6.5 months postpartum
  The outcome is a binary variable, set to 1 if a participant reports using any of the most effective family planning methods as classified by the US CDC at the time of the survey. The subset of the most effective methods includes: implant, IUD, sterilization, injectable, pill, patch, diaphragm, and ring.
Time to take-up of most effective methods | 0-6.5 months postpartum
  This outcome is a continuous time variable, measured in weeks, representing the interval between delivery and first adoption of one of the most effective methods of family planning, as classified by the CDC. This outcome is calculated only for participants who reported using one or more of these most effective methods.
Discussion of FP at any prenatal visit | 3 months postpartum
  The outcome is a binary variable, assigned a value of 1 if a participant reports having had a discussion about family planning with their antenatal care provider at any point during the prenatal period.
Discussion of FP at any postnatal visit | 3 months postpartum
  The outcome is a binary variable, assigned a value of 1 if a participant reports having had a discussion about family planning with health staff at their postnatal care facility at any point during the postnatal period.
Reproductive empowerment: health care provider communication | 3 and 6.5 months postpartum
  The outcome is an average score across 3 items measuring one aspect of reproductive empowerment: health care provider communication (participant reports being able to initiate conversations about using contraception with health care providers, ask health care provider questions about using contraception, and share opinions about using contraception with health care providers.)

OTHER OUTCOMES:
Quality of helpdesk team in counselling on family planning | 6.5 months postpartum
  This outcome is a discrete variable with values ranging from 1 (not helpful at all) to 5 (very helpful), indicating the quality of the helpdesk team's counseling on family planning methods. This outcome is measured only among participants who have interacted with a helpdesk agent.
Quality of message flow on method selection | 6.5 months postpartum
  This outcome is an index with scores ranging from 3 to 15, based on three items with discrete scales measuring the quality of the message flow from the PROMPTS platform regarding method selection. Each item ranges from 1 (not helpful at all) to 5 (very helpful), assessing the usefulness of the messaging platform in: 1) educating about different family planning methods, 2) providing information related to any concerns or issues they had with family planning methods, and 3) assisting in the selection of a family planning method.

CONTACTS AND LOCATIONS:
Overall Officials: Anneka Wickramanayake, MPH, Principal Investigator — Jacaranda Health
Locations (1):
- Jacaranda Health, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No